CLINICAL TRIAL: NCT06030713
Title: Timing of Umbilical Cord Clamping During an Elective Caesarean Delivery and Its Association With Neonatal Gut Microbiome.
Brief Title: Timing of Maternal Antibiotic Prophylaxis During a Cesarean Section and the Early Infant Gut Microbiome
Acronym: CSBabyBiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CS_Baby_Biome_2017/240; NL61493.042.17 (Registry Identifier: ABR); METc 2017.240 (Other: METc)
Record Dates: First submitted 2023-08-25; First posted 2023-09-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Microbial Colonization; Antibiotic Side Effect; Cesarean Section Complications
MeSH Terms: conditions — Communicable Diseases | interventions — Cefazolin

STUDY DESIGN:
Intervention Model Description: Timing of umbilical cord clamping is different in the two arms. One gram of Cefazolin (once, intravenous) will be given to one group of women before skin incision compared to 1g cefazolin given to another group of women after umbilical cord clamping during an elective caesarean section.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cord clamped after antibiotic prophylaxis (Active Comparator): Umbilical cord clamped after 1g of cephazolin
  Interventions: Drug: Cefazolin
- Cord clamped before antibiotic prophylaxis (Experimental): Umbilical cord clamped before 1g of cephazolin
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Cord clamping before or after antibiotic (cefazolin) prophylaxis
  Other Names: DB01327; J01DB04

SUMMARY:
In this study, investigators seek to determine whether the timing of antibiotics given to mothers during an elective C-section affects the composition of their infant's gut microbiome. To do this, a randomized controlled trial (RCT) was carried out with women undergoing elective C-sections. These women were either given antibiotics before the skin incision (AB+) or after the umbilical cord was clamped (AB-).

DETAILED DESCRIPTION:
Rationale: During a caesarean delivery, umbilical cord clamping can occur before or after administering a perioperative prophylactic antibiotic to the mother. If the cord is clamped before the antibiotic administration, this antibiotic cannot reach the infant. Conversely, if the cord is clamped after the antibiotic administration, these maternal antibiotics cross the placenta and enter the infant's circulation. In this study, investigators hypothesize that such antibiotics modify the composition and functionality of the neonatal gut microbiome. A changed neonatal microbiome associates with the onset of asthma, allergies, type 1 diabetes, and obesity later in life. Such a small intervention could influence the future health of the infant significantly.

Objective: The primary aim of this study is to contrast the composition and functionality of the neonatal gut microbiome from mothers given antibiotic prophylaxis before skin incision with the microbiome of neonates from mothers given the antibiotic after umbilical cord clamping during an elective caesarean delivery.

Study design: Randomized controlled trial

Study population: Pregnant women at >38 weeks of gestation undergoing elective caesarean section at the UMCG will be randomized into two groups. The gut microbiome of the neonates from both groups will be analyzed.

Intervention: The timing of umbilical cord clamping differs between the two groups. One gram of Cefazolin (once, intravenous) will be administered to one group before skin incision, while 1g cefazolin will be given to another group after umbilical cord clamping during an elective caesarean section.

Main study parameters/endpoints: The primary endpoint of this study is the variance in the composition and functionality of the neonatal gut microbiome over a year, contrasting neonates from mothers given antibiotic prophylaxis before skin incision with neonates from mothers given the antibiotic after umbilical cord clamping.

ELIGIBILITY:
Inclusion Criteria:

* Females undergoing elective CS at the UMCG
* Gestational age in weeks equal to or above 38 weeks

Exclusion Criteria:

* Cephalosporin allergy
* Exposure to antibiotic agent 2 weeks before CS
* Temperature >37.5 C before CS
* Pre-labour rupture of membranes
* Emergency CS
* No -20 freezer at home
* No command of the Dutch language

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Infant microbial species level differences between two groups | First 6 weeks of life
  Centered log ratio transformed relative abundance differences of bacterial species (relative abundance of > 0.05% and present in at least 2 infants) between two interventional groups
Infant Alpha Diversity differences between two groups | First 6 weeks of life
  Alpha Diversity difference measured by the Shannon Diversity Index of infant microbiome at species level between two interventional groups
Infant Beta Diversity differences between two groups | First 6 weeks of life
  Beta Diversity difference in Aitchison distances between the two intervention groups
Infant Antibiotic Resistance total gene load differences between two groups | First 6 weeks of life
  Infant Antibiotic Resistance total gene load differenced measured in RPKM between the two interventional groups

SECONDARY OUTCOMES:
Number of participants with post c-section maternal wound infection | First 6 weeks of life
  Number of participants with early and late post C-section wound infection in mothers

CONTACTS AND LOCATIONS:
Overall Officials: Trishla Sinha, MD, Principal Investigator — University Medical Center Groningen; Alexandra Zhernakova, MD/PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The sequencing data of the microbiome will be available for other researchers via EGA
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available upon publication
Access Criteria: Must fill in the form that the data will be used for research purposes.